CLINICAL TRIAL: NCT05210647
Title: Analysis of Surgical Outcome of Robotic Surgery Versus Conventional Laparoscopy Surgery. Retrospective Case Control Study in Single Institute.
Brief Title: Robotic Assisted Colon and Rectal Surgery Prognostic and Outcome Analysis
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CE21319A
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-01-27 (Actual); Status verified 2022-01

CONDITIONS: Colorectal Disorders
Keywords: robot, laparopscopy, MIS, surgical outcome, da Vinci Xi,
MeSH Terms: interventions — Robotic Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- conventional laparoscopy surgery: Conventional laparoscopy surgery for colon and rectal disease.
- robot assisted surgery: robotic assisted surgery for colon and rectal disease.
  Interventions: Device: robotic surgery

INTERVENTIONS:
Device: robotic surgery — by da Vinci Xi
  Groups: robot assisted surgery

SUMMARY:
To analysis surgical outcome between robotic and laparoscopy colon and rectal surgery. Retrospective case-control study of single institute.

DETAILED DESCRIPTION:
Microinvasive surgery bring minor pain, faster recovery and comparable oncological outcome. Robotic surgery seems to be superior in precise dissection then before. This study compare robot assisted to laparoscopy surgery in colon and rectal disease. To analysis the surgical outcome and prognostic factors.

ELIGIBILITY:
Inclusion Criteria:

* for colon and rectal disease, using conventional laparoscopy and da Vinci Xi robot system.

Exclusion Criteria:

* emergent operation, combined other open surgery, for non-colorectal disease, carcinomatosis found to be unsuitable for surgery once peritoneum entered, taTME in laparoscopy group and other robot system in robotic surgery group.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From 2019.1.1 to 2022.1.8. Robot surgery team in department of colorectal surgery in TCVGH leaded by Surgeon A and B conducted 142 robot surgery using da Vinci Xi. Meanwhile, they also done 150 conventional laparoscopy surgery. The study compare the surgical outcome and relative prognostic factors between laparoscopy and robotic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2022-01-08 (Actual)

PRIMARY OUTCOMES:
surgical outcomes | 2019.1.1-2022.1.8
  operation time, blood loss, hospital stay, complication rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan